CLINICAL TRIAL: NCT01269320
Title: Natural Soybean-derived Femarelle ®for Patients With Non Alcoholic Fatty Liver Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsors decision
Sponsor: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0172-10-HMO-CTIL
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-08

CONDITIONS: Nash
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — DT56a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Femarelle — Study treatment will consist of Femarelle, two 530mg oral tablets (equivalent to 322 mg of DT56a and 108 mg of Linum Usitatissimum extract each) twice a day for 90 days

SUMMARY:
This is a Single -arm, open-label, before-and after exploratory trial of 90 days of Femarelle ® to improve NAFLD and the metabolic syndrome.

Ingestion of Femarelle will improve non alcoholic steatohepatitis and the metabolic syndrome in patients suffering from these conditions.

Subjects will receive treatment with Femarele 530 mg (1 capsule twice a day) for 90 days and will then be monitored off study treatment for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven NASH
2. If suffering from diabetes may be treated by up to 2 oral medications, with stable doses for 2 months.
3. If participating in sexual activity that could lead to pregnancy, the study volunteer must agree that two reliable methods of contraception will be used simultaneously while receiving the protocol-specified medication and for 1 month after stopping the medication.

   NOTE: Hormonal-based methods alone are not sufficient. At least two of the following methods MUST be used appropriately unless documentation of menopause, sterilization, or azoospermia is present:
   * Condoms (male or female) with or without a spermicidal agent. - Condoms are recommended because their appropriate use is the only contraception method effective for preventing HIV transmission
   * Diaphragm or cervical cap with spermicide
   * IUD
   * Hormonal-based contraception

   Study subjects who are not of reproductive potential (girls who have not reached menarche or women who have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy and/or bilateral oophorectomy are eligible without requiring the use of contraceptives. Written or oral documentation communicated by clinician or clinician's staff is required by one of the following:
   * Physician report/letter
   * Operative report or other source documentation in the patient record (a laboratory report of azoospermia is required to document successful vasectomy)
   * Discharge summary
   * Laboratory report of azoospermia
   * FSH measurement elevated into the menopausal range as established by the reporting laboratory.
4. Ability and willingness of subject or legal guardian/representative to provide informed consent.

Exclusion Criteria:

1. Pregnancy or Breast-Feeding
2. Continuous use of the following medications for more than 3 days within 30 days of study entry:

   * Immunosuppressives
   * Immune modulators
   * Systemic glucocorticoids
   * Anti-neoplastic agents
3. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
4. Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.
5. Surgery within the previous 3 months.
6. Any serious infectious, cardiac, pulmonary, or kidney disease
7. Hypersensitivity to Femarelle ®
8. Malignancy of the uterus or breast
9. Past thromboembolic event

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel